CLINICAL TRIAL: NCT06214676
Title: Detection of Microvascular Changes in Patients With Primary Open Angle Glaucoma by Using Optical Coherence Tomography Angiography
Brief Title: OCTA in Patients With Primary Open-angle Glaucoma
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Yara Ahmed Mohamed, resident doctor at internal ophthalmology department, Assiut University
Other Study IDs: OCTA in glaucoma
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: OCT angiography — Detection of microvascular changes in patients with primary open angle glaucoma by using Optical Coherence Tomography Angiography

SUMMARY:
Is to investigate retinal microvascular changes in primary open angle glaucoma patients using Optical Coherence Tomography Angiography.

DETAILED DESCRIPTION:
Optical coherence tomography angiography (OCT-A) is a non-invasive imaging technique developed to visualize vascular networks in the retina and choroid. It utilizes low-coherence interferometry to measure changes in backscattered signal to differentiate areas of blood flow from areas of static tissue.

OCTA provides both structural and functional (i.e. blood flow) information in tandem. The "corresponding" OCT b-scans can be co-registered with the simultaneous OCT angiograms so the operator is able to scroll through the OCT angiogram like a cube scan. As a result, the precise location of pathology can be viewed on the corresponding OCT b-scans. This makes OCTA a better tool when detecting the exact location of a retinal pathology.

Glaucoma is the first cause of irreversible blindness and represents approximately 15% of all causes of blindness . This makes it a real public health problem. In 2020, glaucoma affected about 80 million people worldwide, with nearly 75% of open-angle glaucoma Primary open-angle glaucoma (POAG) is a chronic, progressive, blinding, irreversible optic neuropathy characterized by damage to the optic nerve head and retinal nerve fibers with subsequent visual field defects ,elevated intraocular pressure (IOP) is a crucial glaucoma risk factor that causes direct damage to RGCs and the optic nerve . Moreover, glaucomatous retinsl ganglion cells loss occurs as well in people with normal IOP, implying mechanisms behind pressure-mediated damage. RGCs death may be due to the reduced blood supply and microvasculature dysfunction may be essential in glaucoma pathogenesis .

One hypothesis is that POAG is categorized by impaired chemical endothelial signaling between both: a) the inner wall Schlemm's canal endothelial cells as well as endothelial cells located in the ciliary body and the posterior longitudinal muscle that helps to set outflow resistance and b) the ocular vascular endothelial cell and underlying luminal smooth muscle for vessels supplying the retinal ganglion cells (RGCs). This hypothesis could explain why POAG occurs across a spectrum of IOP but it does not consider the role systemic endothelial cell dysfunction may play in the disease.

The non-invasive technique of OCT angiography (OCTA) can image and quantify both large vessels and the microvasculature of the optic nerve head (ONH), retina and choroid layers . Using the OCTA technique, reduced vessel density (VD) was observed in the ONH, peripapillary area and macula, predominantly in primary open-angle glaucoma (POAG)

ELIGIBILITY:
Inclusion Criteria:

- clinical diagnosis of Primary open angle glaucoma.

Exclusion Criteria:

* media opacity
* poor fixation due to advanced disease
* associated vascular retinopathy
* chronic uveitis
* optic nerve disease due to other etiologies

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary open angle patients presented to El Nour Eye Center data will be collected by scientifically qualified and trained resident doctors using Optical Coherence Tomography Angiography ( solix)
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
to detect and evaluate microvascular changes in primary open angle glaucoma both qualitatively and quantitatively. | Baseline
  Detection of microvascular changes in patients with Primary open-angle glaucoma